CLINICAL TRIAL: NCT05475093
Title: Evaluation of Impact of Different Micturition Modes on Patients With Medullar Injury of Their Quality of Life and Their Occupations
Brief Title: Impact Evaluation of Different Micturition Modes on Patients With Medullar Injury of Quality of Life and Their Occupations
Acronym: URO-ActSCi
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220265; 2021-A02637-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Medullary Injury; Micturition Disorder
Keywords: Medullary Injury; Micturition modes; Quality of life; Human occupation
MeSH Terms: conditions — Urination Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the study is to analysis the personal determination factors (age, sex, stage of injury, pain, urinary continence and durations of spinal cord injury) and environmental determination factors (need for medical devices, nurse care and adaptation of accommodations) which affect the quality of life and their occupations on patients with medullar injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with spinal cord injury;
* Live at home or in long-term care facility definitively;
* Have one of the following urination modes:

  1. urine with indwelling catheter in place
  2. catheter in suprapubic area
  3. intermittent catheterization by urethra
  4. intermittent catheterization by incontinent cystostomy
  5. sphincterotomy
  6. incontinent stomia (Bricker)

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with medular injury who have their follow-up care in the neuro-urology unit in raymond poincaré hospital, live at home or in long-term care facility definitively.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Quality of life by QUALIVEEN-30 | at baseline
  The questionnaire QUALIVEEN-30 will be used to evaluate the quality of life. It's a reliable tool specially for patients with medullar injury and recommended by the European Association of Urology as Guideline since 2008. The french version is validated.
Model of human occupation | at baseline
  Questionnaire MCREO (french version) will be used to evaluate patients in the occupational aspect.

CONTACTS AND LOCATIONS:
Overall Officials: Alexia EVEN, MD, Principal Investigator — Neuro-Urology Unit, Physical Medicine and Rehabilitation Department, Raymond Poincaré Hospital, APHP; Aurélie -Anna DUBOIS, Study Director — Neuro-Urology Unit, Physical Medicine and Rehabilitation Department, Raymond Poincaré Hospital, APHP
Locations (1):
- Neuro-Urology Unit, Physical Medicine and Rehabilitation Department, Raymond Poincaré Hospital, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No